CLINICAL TRIAL: NCT07197437
Title: Clinical Efficacy of Resin Based Coating Materials for Protecting Dental Root
Brief Title: Efficacy of Universal Bonding Agents as Desensitizers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Hospital of Stomatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKUSSIRB-202273039; PKUSSIRB-202273039 (Other: the Ethical Committee of Peking University School and Hospital of Stomatology); MR-11-22-005868 (Other: https://www.medicalresearch.org.cn)
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Bond Universal (Experimental): Use a microbrush to apply a drop of agent to the sensitive tooth surface for 20 seconds and light cure.
  Interventions: Device: Single Bond Universal as desensitizer
- Hybrid Coat (Active Comparator): Use a coated cotton pellet to apply a drop of agent to the sensitive tooth surface for 20 seconds and light cure.
  Interventions: Device: Hybrid Coat desensitizer

INTERVENTIONS:
Device: Hybrid Coat desensitizer — Dental desensitization treatment
  Arms: Hybrid Coat
Device: Single Bond Universal as desensitizer — Dental desensitization treatment
  Arms: Single Bond Universal

SUMMARY:
The goal of this clinical trial is to learn if the adhesive Single Bond Universal works to treat dentin hypersensitivity in adults. It will also learn about the durability of Single Bond Universal. The main questions it aims to answer are:

Does Single Bond Universal has the function to treat dentin hypersensitivity in adults? Researchers will compare Single Bond Universal to a traditional desensitizer Hybrid Coat to see which one has higher efficiency and longer durability.

Participants will:

Receive the treatment of Single Bond Universal or Hybrid Coat at the first visit.

Visit the clinic at 1, 3, 6, 9, 12 months for follow-up evaluation. Reassess dentin sensitivity at each visit and record in terms of VAS score.

DETAILED DESCRIPTION:
This is a randomized, double-blind and controlled study to include 14 patients with dentin sensitivity. The study is a randomized controlled trial with split mouth control, with symmetrical tooth positions on both sides of the same patient as test and control groups, the test group being the group using the universal bonding agent and the control group being the group using the clinically used desensitizer (Hybrid Coat). Improvement in dentin sensitivity symptoms was the primary outcome indicator observed. Dentin sensitivity was assessed by evaluating the reduction in dentin sensitivity VAS scores at immediately, 1 month, 3 months, 6 months, 9 months and 12 months points after the desensitization treatment. Safety was assessed by evaluating appliance defects and adverse events at the same time points after the desensitization treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥ 18 years who were able to provide written informed consent.
2. Participants confirmed as healthy according to the examiner, without clinically significant diseases that could interfere with study outcomes.
3. Participants with symptoms of dentin hypersensitivity affecting symmetrical teeth on both sides due to gingival recession.
4. Symptomatic teeth without caries, filling materials, or use as abutments for removable partial dentures.

Exclusion Criteria:

1. Individuals with dentin hypersensitivity caused by other factors (e.g., erosion or wedge-shaped defects).
2. Individuals with teeth exhibiting deep periodontal pockets (≥ 4 mm) or with a difference in gingival recession between the two symptomatic teeth of ≥ 1 mm.
3. Individuals who had received treatment or used toothpaste for dentin hypersensitivity within the previous 4 weeks.
4. Individuals who had undergone tooth bleaching or periodontal treatment within the previous 4 weeks.
5. Individuals who had undergone cervical restorative treatment. Individuals who had taken nonsteroidal anti-inflammatory drugs or narcotic analgesics within the previous week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
treatment efficacy of the tooth: the change in VAS score before and after desensitization | from enrollment to the last follow-up (12 months after treatment)
  The severity of dentin sensitivity is assessed using visual analogue scale (VAS) with numbers 0-10 by participants after cold air stimulation. Beforehand, the participants were informed that the 10 cm VAS would be used to assess their pain sensitivity, with 0 indicating no pain and 10 indicating the worst pain. Lower scores on the VAS indicate lower sensitivity. Dentin sensitivity was considered to have improved if the visual pain scale (F-VAS) score decreased by 2 or more points from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Cai, Principal Investigator — Peking University School and Hospital of Stomatology
Locations (1):
- Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The protocol and results will be displayed in a published article. Other dataset containing participants' information cannot be made public according to the requirements of the informed consent form.